CLINICAL TRIAL: NCT03013478
Title: Computer Based Training in CBT in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1607018152; R01DA030369 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment as usual (TAU) (No Intervention): Treatment normally offered at this primary care clinic
- TAU plus CBT4CBT program (Active Comparator): Treatment normally offered at this clinic PLUS 8 weeks of CBT4CBT computerized therapy.
  Interventions: Behavioral: Standard Treatment As Usual (TAU); Behavioral: CBT4CBT program

INTERVENTIONS:
Behavioral: Standard Treatment As Usual (TAU) — Treatment normally offered at this primary care clinic
  Arms: TAU plus CBT4CBT program
Behavioral: CBT4CBT program
  Arms: TAU plus CBT4CBT program

SUMMARY:
To conduct an 8-week randomized trial evaluating the feasibility and efficacy of adding CBT4CBT to treatment as usual in a community based primary care program in a population of 60 individuals who meet current DSM criteria for substance use disorder other than nicotine.

DETAILED DESCRIPTION:
The investigators will conduct an initial evaluation of the computer program as an enhancement of treatment as usual in a community-based primary care clinic. Sixty individuals with a current DSM-IV alcohol or substance use disorder will be randomly assigned to either (1) treatment as usual, or (2) treatment as usual plus exposure to the 'CBT for CBT' program over a period of 8 weeks. Primary outcomes will be retention in treatment and reduction in drug use over 8 weeks. Secondary outcomes include treatment utilization

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older.
* Are applying for outpatient substance abuse treatment
* Meet current DSM-IV criteria for cocaine, marijuana, opioid, alcohol or other stimulant use disorder
* Are sufficiently stable for 8 weeks of outpatient treatment
* Can commit to 8 weeks of treatment and are willing to be randomized to treatment
* Are willing to provide locator information.

Exclusion Criteria:

* Have an untreated bipolar or schizophrenic disorder
* Have a current legal case pending such that incarceration during the 8 week protocol is likely
* Are in need of detoxification from alcohol, opioids or benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
retention in treatment | 0 - 8 weeks
  subjects returning for treatment at primary care unit and completing CBT4CBT program for those assigned
reduction in drug use | 0 - 8 weeks
  Using urine and breathalyzer screening for negative drug and alcohol testing

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital St Raphael's Campus, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tetrault JM, Holt SR, Cavallo DA, O'Connor PG, Gordon MA, Corvino JK, Nich C, Carroll KM. Computerized Cognitive Behavioral Therapy for Substance Use Disorders in a Specialized Primary Care Practice: A Randomized Feasibility Trial to Address the RT Component of SBIRT. J Addict Med. 2020 Dec;14(6):e303-e309. doi: 10.1097/ADM.0000000000000663. PMID 32371660